CLINICAL TRIAL: NCT00840203
Title: A Study to Evaluate the Relative Bioavailability of Two Mesalamine 4 gm/60 mL Rectal Enema Formulations
Brief Title: Mesalamine 4 gm/60 mL Rectal Enema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10336014
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamine (Experimental): Mesalamine 4gm/60mL Rectal Enema (test) dosed in first period followed by Rowasa® 4gm/60mL Rectal Enema (reference) dosed in second period
  Interventions: Drug: Mesalamine 4 gm/60 mL Rectal Enema
- Rowasa® (Active Comparator): Rowasa® 4gm/60mL Rectal Enema (reference) dosed in first period followed by Mesalamine 4gm/60mL Rectal Enema (test) dosed in second period
  Interventions: Drug: Rowasa® 4 gm/60 mL Rectal Enema

INTERVENTIONS:
Drug: Rowasa® 4 gm/60 mL Rectal Enema — 1 x 4 gm/60 mL, single-dose
  Arms: Rowasa®
Drug: Mesalamine 4 gm/60 mL Rectal Enema — 1 x 4 gm/60 mL, single-dose
  Arms: Mesalamine

SUMMARY:
The objective of this study is to evaluate the relative bioavailability of the test formulation of mesalamine suspension rectal enema with the already marketed reference formulation Rowasa® in healthy, adult subjects.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older, with a body mass index (BMI) of 30 or less.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed informed consent form, which meets all criteria of current FDA regulations.
* If female and of child bearing potential prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g. condom, IUD, hormonal contraceptives).

Exclusion Criteria:

* If female pregnant, lactating, or likely to become pregnant during the study.
* History of allergy or sensitivity to mesalamine or other salicylic drugs (e.g. aspirin, sulfasalazine) or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Colitis, hemorrhoids, anal fissures, or other disease of the anus, rectum or colon.
* Significant history or current evidence of chronic infections disease, system disorder or organ disorder.
* History of psychiatric disorders occuring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs (other than contraceptives).
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to dosing.
* Positive test for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Positive serum pregnancy test at screening.
* Unable or unwilling to tolerate multiple venipunctures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-05; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Ann Kennedy, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesalamine (Test) First: Mesalamine 4gm/60mL Rectal Enema (test) dosed in first period followed by Rowasa® 4gm/60mL Rectal Enema (reference) dosed in second period
- Rowasa® (Reference) First: Rowasa® 4gm/60mL Rectal Enema (reference) dosed in first period followed by Mesalamine 4gm/60mL Rectal Enema (test) dosed in second period
Period: First Intervention
Arm/Group | Mesalamine (Test) First | Rowasa® (Reference) First
Started | 37 | 35
Completed | 36 | 34
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Washout
Arm/Group | Mesalamine (Test) First | Rowasa® (Reference) First
Started | 36 | 34
Completed | 35 | 34
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Mesalamine (Test) First | Rowasa® (Reference) First
Started | 35 | 34
Completed | 35 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalamine (Test) First | Rowasa® (Reference) First | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 35 | 72
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 23 | 23 | 46
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 18 | 17 | 35
  Black | 17 | 16 | 33
  Hispanic | 0 | 1 | 1
  Biracial | 0 | 1 | 1
  Asian | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Mesalamine: Mesalamine 4gm/60mL Rectal Enema (test) dosed in either period
- Rowasa®: Rowasa® 4gm/60mL Rectal Enema (reference) dosed in either period
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 69 | 69
ng/mL | 1451.739 (718.488) | 1500.290 (778.674)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — Using the General Linear Model (GLM) procedure of SAS the bioequivalence of the test and reference products will be evaluated using average bioequivalence methodology for non-replicate crossover study design; Geometric Test/Ref Ratio x 100 = 97.6, 90% CI [88.6 to 107] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 48 hour period
Population: AUC0-inf was not able to be estimated for all completing subjects
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 52 | 56
ng*h/mL | 24458.932 (16649.166) | 26862.895 (21419.555)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 97.3, 90% CI [82.8 to 114] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 69 | 69
ng*h/mL | 21543.597 (15674.400) | 22911.830 (15380.728)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 94.0, 90% CI [83.0 to 107] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Secondary Outcome: Cmax - Maximum Observed Concentration
Description: Cmax results for N-Acetylmesalamine metabolite
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 69 | 69
ng/mL | 2274.652 (934.469) | 2284.884 (857.980)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 98.3, 90% CI [91.5 to 106] — Metabolite results presented for informational purposes only

5. Secondary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: AUC0-inf results for N-Acetylmesalamine metabolite
Time Frame: Blood samples collected over 48 hour period
Population: AUC0-inf was not able to be estimated for all completing subjects
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 60 | 58
ng*h/mL | 46564.373 (29109.234) | 49692.278 (32182.649)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 97.6, 90% CI [86.7 to 110] — Metabolite results presented for informational purposes only

6. Secondary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: AUC0-t results for N-Acetylmesalamine metabolite
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mesalamine | Rowasa®
Number analyzed (Participants) | 69 | 69
ng*h/mL | 40873.915 (25272.348) | 42644.677 (24335.847)
Statistical Analysis 1: Comparison: Mesalamine vs Rowasa®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 95.6, 90% CI [86.1 to 106] — Metabolite results presented for informational purposes only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.